CLINICAL TRIAL: NCT00663507
Title: Kidney Transplantation in Patients With Sickle Cell Disease
Status: Terminated | Type: Observational
Why Stopped: Only 1 patient was enrolled. No funding, small number of eligible patients so would not achieve statistical power.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nicole Turgeon MD, Assistant Professor, Emory University
Other Study IDs: IRB00004914
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Immunosuppression; Organ & Tissue Transplantation; Transplantation Immunology
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 100 mLs of whole blood will be collected at designated time points. Baseline, and at 1,3,6,9,12,18 and 24 months post-transplant
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research is to better characterize the components and mechanisms of the immune systems of persons with sickle cell disease who have had a kidney transplant and are immunosuppressed. If we can improve our scientific understanding of the fundamental mechanisms involved in patient outcomes, we can potentially maximize the benefits that we seek from transplantation in sickle cell patients with end stage renal disease.

DETAILED DESCRIPTION:
Sickle cell disease is a common disease in the African-American population. In sickle cell disease red blood cells are abnormal in shape and can damage organs. In particular, patients with sickle cell disease can have damage to the kidneys, resulting in renal failure. The number of patients developing renal failure with sickle cell disease is unknown. This is largely due to the high mortality of patients with sickle cell disease and renal failure.

There are two types of renal replacement therapy available to patients with sickle cell disease- dialysis and kidney transplantation. The best form of renal replacement therapy has not been determined for patients with sickle cell disease and renal failure. There have been approximately 190 renal transplants performed in the United States since 1988 in patients with sickle cell disease. Patients do well, but do not survive as long as patients with other causes of renal failure. It appears that patients with sickle cell disease who meet the criteria for kidney transplantation may derive a benefit from transplantation rather than undergoing dialysis.

We are performing this study to follow patients with sickle cell disease who have received a renal transplant. We hope to learn the best way to manage patients with sickle cell disease to improve both survival of the transplanted kidney and the patients.

In addition, we are studying the immune system and how it responds to receiving a kidney transplant in sickle cell patients. We hope the information we learn about the immune system will allow us to prevent injury to the new kidney transplant and allow for better outcomes in sickle cell patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 65 years of age
2. Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study.
3. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and must not be breast-feeding.
4. Patients must be diagnosed with Sickle Cell Disease (SS phenotype)

Exclusion Criteria:

1. Patients with any prior organ transplant or multi-organ transplant recipients.
2. Patients with evidence of an active systemic infection requiring the continued use of antibiotics, evidence of an HIV infection, or the presence of a chronic active hepatitis B or C.
3. Patients with history of malignancy in the last 5 years (except successfully treated localized non-melanotic skin cancer)
4. Patients with active illegal drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of sickle cell disease (SS type) with end stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
No measure applied | 05/08/2008-6/05/2009
  One 12 month participant, with no actions. One subject was a screen failure due to hepatitis C.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Turgeon, M.D., Principal Investigator — Emory University
Locations (1):
- Mason Outpatient Tranplant Clinic Emory University, Atlanta, Georgia, United States